CLINICAL TRIAL: NCT04636593
Title: Almonertinib With Concurrent Radiotherapy in The Treatment of Unresectable, Stage Ⅲ Non-small-cell Lung Cancer Harboring EGFR Mutations: A PhaseⅡCohort Study
Brief Title: A Phase 2 Trial of Almonertinib With Concurrent Radiotherapy in The Treatment of Local Advanced EGFR-mutant NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First People's Hospital of Hangzhou (Other)
Collaborators: Hangzhou Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AlmonTRT
Record Dates: First submitted 2020-11-15; First posted 2020-11-19 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Non Small Cell Lung Cancer; Stage III NSCLC; EGFR Activating Mutation
Keywords: radiotherapy; radiation pneumonitis; almonertinib; lung cancer; EGFR-TKI
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Radiation Pneumonitis; Lung Neoplasms | interventions — aumolertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Induction group (Experimental): If the lung V20 of initial radiation plan is equal to or more than 28%, then the patient will receive 2 months almonertinib before concurrent thoracic radiotherapy
  Interventions: Drug: Almonertinib
- Concurrent group (Experimental): If the lung V20 of initial radiation plan is less than 28%, then the patient will receive concurrent thoracic radiotherapy with almonertinib.
  Interventions: Drug: Almonertinib

INTERVENTIONS:
Drug: Almonertinib — All enrolled patients underwent positioning CT scans before the initial treatment, a radiotherapy plan was made for each patient, and the lung V20 of each patient was calculated. Patients with lung V20 ≥ 28% were enrolled in group A: Almonertinib induction therapy was given for 2 months firstly, followed by Almonertinib combined with radiotherapy; patients with lung V20<28% were enrolled in group B: Almonertinib was synchronized with radiotherapy initially.
  Other Names: Thoracic Radiotherapy

SUMMARY:
Previous clinical studies showed there is a potential value of EGFR-TKI in local advanced EGFR-mutant NSCLC, while the risk of radiation pneumonia in combination of EGFR-TKI with thoracic radiotherapy is unknown. This study aims to explore the safety and efficacy of concurrent almonertinib, a new third-generation EGFR-TKI drug, with radiotherapy in local advanced EGFR-mutant NSCLC patients.

DETAILED DESCRIPTION:
Doublet platinum-based therapy combined with radiotherapy remains the standard treatment for first-line management of unresectable stage III NSCLC patients, regardless of the EGFR mutation status. But the 5-year survival rate is not satisfying. Previous clinical studies showed there is a potential value but also a high risk of radiation pneumonia in treatment regimens of combination TKI with radiotherapy. This study intends to explore the safety and efficacy of concurrent almonertinib, a new third-generation EGFR-TKI drug, with radiotherapy in EGFR-sensitive mutated locally advanced NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed histologically or pathologically as non-small cell lung cancer;
* According to the eighth edition of the 2015 IASLC international lung cancer staging, imaging staging assessed as inoperable stage III patients (according to the eighth edition of the 2015 IASLC international lung cancer staging);
* Blood or tissue EGFR detection is Exon 19 deletion or L858R mutation;
* Have not received systemic anti-tumor therapy;
* FEV1>0.75L;
* Age ≥ 18 years old;
* ECOG PS score ≤ 2;
* Estimated survival period ≥ 6 months;
* Women must undergo surgical sterilization, post-menopausal, or take contraceptive measures during the treatment period and within 3 months after the end;
* Sign the informed consent form.

Exclusion Criteria:

* Previously received other anti-tumor treatment, including almonertinib or other EGFR-TKI drugs;
* Contraindications for radiotherapy such as uncontrolled systemic lupus erythematosus, scleroderma or other connective tissue diseases;
* Other malignant tumors within 5 years (except for non-melanoma skin cancer and cervical cancer);
* Any medical or non-medical reasons prevent the patient from continuing to participate in the research;
* It is expected that the patient will not be able to comply with the research procedures, restrictions and requirements, and researchers determine that the patient is not suitable for participating in the trial;
* Currently receiving (or unable to stop using it before receiving the first dose of study treatment) drugs or herbal supplements known to be potent inducers of CYP3A4 (at least 3 weeks ago);
* The patient is taking any drugs that prolong the QT interval, and the drug cannot be stopped before the treatment of almonertinib;
* Patients with lung V20 > 28% even after two-month almonertinib treatment.
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
RP(≥3) | 6 months
  incidence of radiation pneumonitis (≥ grade 3) within 6 month after Radiotherapy

SECONDARY OUTCOMES:
LCR | 1 years
  local control rate
PFS | 2 years
  progression-free survival (PFS) defines as intervals from treatment to disease progression or death
OS | 2 years
  overall survival (OS) intervals from treatment to death or last follow-uo

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou Cancer hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu L, Zou C, Zhang Z, Wang J, Yang L, Rao C, Yang Z, Liang J, Xia B, Shenglin MA. Thoracic radiotherapy and concurrent almonertinib for unresectable stage III EGFR-mutated non-small-cell lung cancer: a phase 2 study. BMC Cancer. 2021 May 7;21(1):511. doi: 10.1186/s12885-021-08266-w. PMID 33962566